CLINICAL TRIAL: NCT01543633
Title: Electroencephalogram Studies of Induction and Recovery From Propofol Induced General Anesthesia
Brief Title: EEG Studies of Induction and Recovery From Propofol Induced General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Emery Brown, Emery N. Brown, M.D., Ph.D., Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2005P001549; 5DP1OD003646 (NIH)
Record Dates: First submitted 2012-02-16; First posted 2012-03-05 (Estimated); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Brain Activity Under Sedation
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active Study Arm (Experimental): Subjects recruited into this study will be required to undergo a base MRI scan of the brain. On a separate day propofol will be administered with concurrent EEG while subjects respond to stimuli.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol will be infused using a computer controlled delivery system running the program STANPUMP. Loss of consciousness will be defined as loss of response to auditory stimulus (button press).

SUMMARY:
The purpose of this study is to investigate how the commonly used anesthetic drug propofol works in the brain to produce loss of consciousness. While under general anesthesia your brain waves will be measured using electroencephalogram (EEG). On a separate day, the patient's brain will be imaged using magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking male and female volunteers, ages 18-36 with normal body weight.
* American Society of Anesthesiologists (ASA) physical status I

Exclusion Criteria:

* History of head trauma
* Surgical aneurysm clips
* Cardiac pacemaker
* Prosthetic heart valve
* Neurostimulator
* Implanted pumps
* Cochlear implants
* Metal rods, plates
* Screws
* Intrauterine device
* Hearing aid
* Dentures (which might create NMR artifacts)
* Metal injury to eyes

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2005-08; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emery N Brown, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects with abnormal cardiological abnormality, failure of the hearing test, abnormal ECG reading, and other medical conditions were excluded. Ten subjects also voluntarily withdrawn consent due to scheduling conflicts.
Period: Overall Study
Arm/Group | Active Study Arm
Started | 36
Completed | 17
Not Completed | 19

BASELINE CHARACTERISTICS:
Arm/Group | Active Study Arm
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: Years] | 27 [18 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: EEG Power in Alpha, Slow, and Delta Bands
Description: We used EEG measurements to study the dynamics of loss of consciousness, auditory processing, sensation, and memory under general anesthesia induced with propofol. The EEG data in each of the three specific aims will be analyzed using spectral methods, source localization, and event-related potentials. Through spectral analysis, EEG power (in decibels) in alpha, slow, and delta bands are measured.
Time Frame: 11 hours
Measure: Median (95% Confidence Interval); unit: Power of alpha band (decibels)
Arm/Group | Active Study Arm
Number analyzed (Participants) | 17
Power of alpha band (decibels)
  Alpha Band Power | 10 [8 to 12]
  Slow Band Power | 0.55 [0.1 to 1]
  Delta Band Power | 2.5 [1 to 4]

ADVERSE EVENTS:
Time Frame: 24 hours. The day after completion of the anesthesia portion of the study, a follow-up call will be made by the study subject's dedicated anesthesiologist to ensure that the study subject has fully recovered and has no health concerns or problems related to the study.
Description: The definition of adverse event and/or serious adverse event does not differ from the clinical trials.gov definitions.
  Note that the study was stopped if the blood pressure fell out of the range of 20% of the baseline values of end-tidal CO2, pulse oximetry levels, O2 saturation, and blood pressure. The study was also aborted if there is a problem with the placement of the intra-arterial or intravenous catheter.
Arm/Group | Active Study Arm
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT01543633/Prot_SAP_000.pdf